CLINICAL TRIAL: NCT03179683
Title: Radiographic Evaluation of Low Level Laser Therapy Enhanced Maxillary Sinus Augmentation With Simultaneous Implant Placement
Brief Title: Effect of Low Level Laser Teraphy on Bone Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ugur GULSEN (Other)
Responsible Party: Sponsor-Investigator, Ugur GULSEN, Principal investigator, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 824-02/9-8/97
Record Dates: First submitted 2017-05-29; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Alveolar Ridge Augmentation
Keywords: aluminum step-wedge; demineralized bone matrix; dental implant; digital densitometry; low level laser therapy; maxillary sinus augmentation.

STUDY DESIGN:
Intervention Model Description: The study was planned as randomized controlled split-mouth clinical study. Bilateral sinus bone augmentation and dental implant surgeries were done simultaneously. Low level laser therapy (LLLT) was (λ= 630-660 nm, 25 mw / cm², 6 mins) applied for just one operation side at first, third, fifth and seventh days. Treatment side were randomly selected by another surgeon who applied LLLT and no treatment were applied to other group(control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diode laser application (Active Comparator): An 630-660 nm aluminum gallium indium phosphide (AlGalnP) laser device (Scorpion Dental Optima Model 405-7A; Optica Laser, Sofia, Bulgaria) was used immediately after surgery, third day, fifth day and seventh day only for one operation side (treatment group)
  Interventions: Device: Diode laser application
- No application (No Intervention): no treatment were aplied

INTERVENTIONS:
Device: Diode laser application — an 630-660 nm aluminum gallium indium phosphide (AlGalnP) laser device (Scorpion Dental Optima Model 405-7A; Optica Laser, Sofia, Bulgaria) was used immediately after surgery, third day, fifth day and seventh day only for one operation side. Treatment side were randomly selected by another surgeon who applied LLLT. Tissue was irradiated at 25mW power for total six minutes, two minutes for each point (buccal, palatal, crestal). 72J /cm2 energy density was deposited in one session.
  Arms: Diode laser application

SUMMARY:
This randomized controlled split-mouth clinical trial study was designed to evaluate the effects of low-level laser therapy on bone healing in patients with bilateral sinus lifting and simultaneous dental implant application.

Maxillary posterior partially edentulous or totally edentulous twelve patients who need bilateral sinus bone augmentation were included in this study. Sinus bone augmentation and dental implant surgeries were done simultaneously. Low level laser therapy (LLLT) was (λ= 630-660 nm, 25 mw / cm², 6 mins) applied for just one operation side at first, third, fifth and seventh days. Treatment side were randomly selected by another surgeon who applied LLLT. Panoramic radiographs were taken at the first, third and sixth months using aluminum step-wedge technique. Optic Density analyses were performed using Cardinal Health Digital Densitometer (Fluke Biomedical 07-443) with 1mm diameter. Digital densitometric results were obtained as equivalent aluminum thickness for each radiograph. These data were used to evaluate changes in optical bone densitometry and compare the LLLT applied side and control side for each patient.

DETAILED DESCRIPTION:
Twelve patients were included to this study who required a bilateral sinus floor augmentation for implant-prosthetic rehabilitation. Nine patients were bilaterally free-end partial edentulous and three patients were totally edentulous with residual alveolar height between 3-6 mm. All patients required bilateral sinus augmentation with simultaneous implant placement.

Patients who have maxillary sinus pathology, previous history of chronic sinus infection, smoking more than ten cigarettes per day, any systemic disease interfere with the surgical procedure were excluded from study.

The study protocol was conducted by Ankara University Dentistry Faculty Research Ethics Committee. All patients were informed about the treatment procedure and all patients gave written consent for participation.

Surgical Protocol Bilateral sinus augmentation and simultaneous implant placement were performed in one appointment with same surgical protocol. All surgical procedures performed under local anesthesia (Ultracain D-S Forte; Sanofi-Aventis, Istanbul, Turkey). After elevation of mucoperiosteal flap a hinge door osteotomy was performed on the lateral wall of the maxillary sinus with a round diamond bur under saline solution irrigation. Schneiderian membrane was carefully detached from inferior and lateral walls of the sinus until creating enough space for placement of bone grafts. Implant osteotomies were performed and DBM putty bone graft (DynaGraft bone putty, Keystone Dental, Burlington, Mass) were placed medial, posterior and anterior side of implant sockets. Implants (Touareg S, Adin, Afula, Israel) were inserted into the osteotomy site after sufficient grafting. Access window filled with bone graft after implant placement. Membrane was not used over access window. 3/0 silk suture were used for closure of the flap. Antibiotic (amoxicillin thrice per day), analgesic (naproxen sodium, 2 twice per day) and mouthwash (isotonic saline twice per day) were prescribed for postoperative management. The patients were advised to have a soft diet and to avoid sneezing until two weeks. Sutures were removed one-week after surgery. No complications occurred during surgery. All surgical wounds healed uneventfully.

Low Level Laser Therapy Protocol In this study, an 630-660 nm aluminum gallium indium phosphide (AlGalnP) laser device (Scorpion Dental Optima Model 405-7A; Optica Laser, Sofia, Bulgaria) was used immediately after surgery, third day, fifth day and seventh day only for one operation side. Treatment side were randomly selected by another surgeon who applied LLLT. Tissue was irradiated at 25mW power for total six minutes, two minutes for each point (buccal, palatal, crestal). 72J /cm2 energy density was deposited in one session.

Radiological Evaluation Aluminum Step-Wedge and Radiographic Assessment Aluminum step-wedge was used as the reference material in densitometric evaluation of the conventional radiographs. The aluminum wedges were prepared using 99,7% pure aluminum plates, the dimensions of the plates were 1 mm in width and 2, 4, 6, 8, 10, 12 mm in length. Prepared six aluminum plates were sticked in a row and a stair-like aluminum wedge had acquired.

Prepared aluminum step-wedges were located in a fixed place (lower left corner) in the film cassettes in order to maintain the calibration and standardization of the radiographs. Special care was taken to avoid the superposition of the hyoid bone and other bony structures with the step-wedge.

In this research, all radiographic assessments were made using panoramic radiographs. The radiographic assessments were done by the same radiology technician from the Oral Diagnosis and Radiology department of Ankara University. Mediphot X-O/RP, sens: green, 15x30 panoramic radiographs were used in this research.

All radiographs were taken with 80 kVp, 12 mA, 2.5 mm Al total filtrated "PM 2002 CC Proline" panoramic radiography device using the same kV and mA values. Radiographic film processing was made in automatic radiograph processing devices, Velopex and Extra-XE.

Four panoramic radiographs were taken from each patient, which were preoperative and postoperative on first., third and sixth months.

Densitometric Assessment Densitometrical analysis was performed on forty-eight radiographs which were taken preoperatively and on postoperative first, third and sixth. Months in this research. Densitometric assessments of the radiographs were made in Medical Physics department of the Ankara University Nuclear Sciences Institute. Cardinal Health Digital Densitometer (Fluke Biomedical 07-443) with 1 mm diameter used in optic density measurement. Results were read and recorded immediately from the devices screen.

Densitometric measurement was repeated three times in each radiograph and an average was acquired, the used spots were every step of the step-wedge and the augmented sinus areas.

Aluminum equivalent thickness of the augmented sinus areas were identified. With this information, the mineralization levels of the graft materials on the radiographs were identified and acquired results were assessed statistically.

Statistical Assessment The Shapiro-Wilk test was used to determine whether the data were normally distributed. The Friedman test was used for four time points in two groups. In cases of significant differences among measurements, the Bonferroni-adjusted Wilcoxon signed-rank test was used as post hoc analysis. Additionally, the Bonferroni-adjusted Wilcoxon signed-rank test (paired observations) was used to compare the two groups in the same time points. All tests were performed using statistical software (SPSS Inc., version 19.0, Chicago, IL, USA). The median with min-max values were calculated for each parameter as the statistical unit. P < 0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Twelve patients were included to this study who required a bilateral sinus floor augmentation for implant-prosthetic rehabilitation. Nine patients were bilaterally free-end partial edentulous and three patients were totally edentulous with residual alveolar height between 3-6 mm. All patients required bilateral sinus augmentation with simultaneous implant placement.

Exclusion Criteria:

Patients who have maxillary sinus pathology, previous history of chronic sinus infection, smoking more than ten cigarettes per day, any systemic disease interfere with the surgical procedure were excluded from study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Bone density analysis | Change from Baseline in Bone Density at 6 months
  Panoramic radiographs were taken using with aluminum step-wedge technique. These images were used to evaluate changes in optical bone densitometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur GULSEN, Principal Investigator — Bulent Ecevit University

IPD SHARING:
Plan to Share IPD: No